CLINICAL TRIAL: NCT05162729
Title: Working Memory Training for Preschoolers at Risk of ADHD and Training Effects on Time Perception, ADHD Symptoms, and Academic Performance
Brief Title: Working Memory and Social-emotional Training for Preschoolers at Risk of ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kathy Shum, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA210224
Record Dates: First submitted 2021-11-02; First posted 2021-12-17 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: ADHD; Time Perception Altered; Working Memory; Social Skills
Keywords: preschool; ADHD; working memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Social Skills

STUDY DESIGN:
Intervention Model Description: Intervention group: receive 5 weeks working memory online training, three times per week, each lasts 15 minutes.
  Active control group: receive 5 weeks social-emotional online training, three times per week, each lasts 15 minutes.
  Control group: no training
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly allocated into groups. Assessors do not know about which group participants were allocated in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Working memory intervention group (Experimental): Receive game-like working memory online training for 5 weeks, 3 times per week, each lasting for15 minutes.
  Interventions: Behavioral: Game-like online working memory training
- Social emotional intervention group (Active Comparator): Receive game-like social-emotional online training for 5 weeks, 3 times per week, each lasting for 15 minutes.
  Interventions: Behavioral: Game-like online social emotional training
- Control group (No Intervention): Receive no training

INTERVENTIONS:
Behavioral: Game-like online working memory training — Participants in the WM group will be receiving two types of WM training tasks (two mini-games) in each session. Half of the training time will be spent on playing a game that requires visual-spatial WM, and the other half of the training time will be spent on playing a game that demands verbal WM. In both the games, the participant is asked to remember the pictures or audios (numbers) presented, and then recall them and select them on the screen.
  Arms: Working memory intervention group
Behavioral: Game-like online social emotional training — Participants in the SE group will be also receiving two types of SE training tasks in each session, to match with the ones in the WM training. There are two mini-games for training.
  To match with the spatial-visual WM training, participants in the SE group will be asked to first look at a picture that depicts a daily social scenario (i.e., a child who fell down and hurt himself), and then to choose an emotion that the child in the picture may feel from four options of facial emotions displayed on the screen. The other mini-game, with the aim to match with the auditory WM training, will first tell a short story of a social scenario (i.e. "David accidentally fell down and got hurt), and then will ask the child to choose the emotion that the character in the story may feel from the four options displayed on the screen. Each mini game lasts for about 7 minutes in each training session.
  Arms: Social emotional intervention group

SUMMARY:
The study aims to explore the effectiveness of working memory training and social emotional training for young children with ADHD in Hong Kong. This study will contribute to the current understanding of the alternative treatments for ADHD, and hopefully help to mobilize more resources to be dedicated to the support of children with ADHD. The programme includes the following components:

Children participating in this study will be randomly allocated into experimental group - recieving working memory training, active control group - receiving social-emotional training, and waitlist control group. All participants will complete a 5-week online training using a digital device at home, three times a week, each training session lasts for about 15 minutes.

Moreover, children's cognitive abilities and academic performance will be assessed prior to the intervention, and immediately after the 5-week training. Each assessment session lasts for about 45 minutes. Parents will also be asked to fill out a questionnaire on children's behaviours at home and school prior to and after the 5-week program. It takes about no more than 10 minutes. All assessments will be conducted at the laboratory at the University of Hong Kong.

Children's working memory, time perception, ADHD symptoms, and early academic performance will be measured before and after training, and the between-group performance will be compared to examine the training effects.

ELIGIBILITY:
Inclusion Criteria:

* children aged 4-6 years old
* with psychiatrist or psychologist diagnosis of ADHD according to the DSM-5 manual or other clinical diagnosis criteria;
* or as indicated by the ratings of Swanson, Nolan and Pelham Parent Rating Scale (SNAP-IV; Chinese version);
* with normal IQ (above 80), which enable them to understand the materials delivered in the training program;
* children either not taking any medication or taking a stable dosage of medication for ADHD for at least 3 months prior to the study enrollment and will not be taking the medication during the training and post-assessment period.

Exclusion Criteria:

* inability to comprehend Cantonese, with comorbid disorders (i.e. autism, conduct/behavioural problems),
* with medical or other mental health condition
* with IQ below 80
* with physical and motor disabilities that restrain them from completing the tasks.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
verbal working memory (CMS- digit span) | 5 weeks, immediately after the intervention
  The number subtest from the Children Memory Scale (Cohen, 1997) was used to measure children's verbal working memory. The Numbers subtest included both digit span forward and backward tasks, for which the children were asked to recall digit sequences presented verbally in increasing length, either in the same order for Numbers Forward or in the reverse order for Numbers Backward. The total score was the sum of the scores for the forward and backward tasks.The raw score scale ranges from 0 to 30. A higher score indicates a better verbal working memory.
verbal working memory(CMS-digit span) | before the intervention
  The number subtest from the Children Memory Scale (Cohen, 1997) was used to measure children's verbal working memory. The Numbers subtest included both digit span forward and backward tasks, for which the children were asked to recall digit sequences presented verbally in increasing length, either in the same order for Numbers Forward or in the reverse order for Numbers Backward. The total score was the sum of the scores for the forward and backward tasks.The raw score scale ranges from 0 to 30. A higher score indicates a better verbal working memory.
non-verbal working memory(CMS - picture location) | 5 weeks, immediately after the intervention
  The picture location subtest from the Children Memory Scale (Cohen, 1997) was used to test participants' non-verbal working memory. Children were asked to look at pictures on a page for 2 seconds and to recall and indicate the pictures' locations by putting chips on the right places that matched the positions of the pictures showed. A score was given when the participant successfully matched the correct position of a picture.The raw score scale ranges from 0 to 30. A higher score indicates a better nonverbal working memory.
nonverbal working memory(CMS - picture location) | before the intervention
  The picture location subtest from the Children Memory Scale (Cohen, 1997) was used to test participants' non-verbal working memory. Children were asked to look at pictures on a page for 2 seconds and to recall and indicate the pictures' locations by putting chips on the right places that matched the positions of the pictures showed. A score was given when the participant successfully matched the correct position of a picture. The raw score scale ranges from 0 to 30. A higher score indicates a better nonverbal working memory.
Time perception: time discrimination | before the intervention
  A computerized task that examined participants' abilities in discriminating discrepancy between different durations of time (Gooch et al., 2011). A threealternative forced-choice (oddball) paradigm was used. On each trial, the child heard three 1000Hz tones, two of which were 1200ms long and a roving target which was at a different length (400ms, 700ms, and 1100ms - each repeated nine times). The child was required to choose which interval was "different" from the other two. Six easy trials of 100ms comparing with 1200ms were incorporated randomly during the experiment to evaluate the attention level of the participants.
Time perception: time discrimination | 5 weeks, immediately after the intervention
  A computerized task that examined participants' abilities in discriminating discrepancy between different durations of time (Gooch et al., 2011). A threealternative forced-choice (oddball) paradigm was used. On each trial, the child heard three 1000Hz tones, two of which were 1200ms long and a roving target which was at a different length (400ms, 700ms, and 1100ms - each repeated nine times). The child was required to choose which interval was "different" from the other two. Six easy trials of 100ms comparing with 1200ms were incorporated randomly during the experiment to evaluate the attention level of the participants.
Time perception: time reproduction | before the intervention
  A computerized lightbulb game was used to measure participants' abilities in recognizing and producing a designated period. The task was adapted from a similar task developed by Gooch and colleagues (2011). It was presented in a computer-game-like format where the child was asked to look at the red lightbulb that would appear on the screen and remember how long it had been left on (3s, 5s, 6s, 9s, 12s, and 15s). After, the child was asked to reproduce for the same length of duration. Immediately following this presentation the screen went blank and the participant was asked to "turn the yellow lightbulb on and leave it on" (use "ENTER" to turn on) for the same amount of time as it had been for the red lightbulb, and then use "SPACE" to turn off the light. Each target duration is presented twice in a randomized order for a total of 12 trials.
Time perception: time reproduction | 5 weeks, immediately after the intervention
  A computerized lightbulb game was used to measure participants' abilities in recognizing and producing a designated period. The task was adapted from a similar task developed by Gooch and colleagues (2011). It was presented in a computer-game-like format where the child was asked to look at the red lightbulb that would appear on the screen and remember how long it had been left on (3s, 5s, 6s, 9s, 12s, and 15s). After, the child was asked to reproduce for the same length of duration. Immediately following this presentation the screen went blank and the participant was asked to "turn the yellow lightbulb on and leave it on" (use "ENTER" to turn on) for the same amount of time as it had been for the red lightbulb, and then use "SPACE" to turn off the light. Each target duration is presented twice in a randomized order for a total of 12 trials.
Time perception: time production | before the intervention
  Subjects were required to indicate the end of 3, 5, 12, and 20-s intervals (each produced twice) by saying "STOP" to indicate the end of the temporal duration.
Time perception: time production | 5 weeks, immediately after the intervention
  Subjects were required to indicate the end of 3, 5, 12, and 20-s intervals (each produced twice) by saying "STOP" to indicate the end of the temporal duration.
Emotion situation knowledge measures. | before the intervention
  This task was developed by Garner et al. (1994) to measure children's ability to infer emotions from situational cues, and similar tasks have been used among preschoolers (Beaudoin et al. 2020; Gallant et al. 2020). Social situations commonly encountered by children were presented in pictures, with the facial expressions of the target characters left out (i.e., blank faces were shown). The children were asked to identify the feeling of the target character by either naming the emotion or pointing to the corresponding facial expression out of four options (happy, sad, angry, and afraid) given on the stimulus sheet. There were two sample items followed by 13 test items.
Emotion situation knowledge measures. | 5 weeks, immediately after the intervention
  This task was developed by Garner et al. (1994) to measure children's ability to infer emotions from situational cues, and similar tasks have been used among preschoolers (Beaudoin et al. 2020; Gallant et al. 2020). Social situations commonly encountered by children were presented in pictures, with the facial expressions of the target characters left out (i.e., blank faces were shown). The children were asked to identify the feeling of the target character by either naming the emotion or pointing to the corresponding facial expression out of four options (happy, sad, angry, and afraid) given on the stimulus sheet. There were two sample items followed by 13 test items.
Theory of mind (ToM) | before intervention
  Children's ToM will be measured by the ToM scale developed by Wellman and Liu (2004). The seven-item scale was designed for the experimental to adminster in order according to the difficulty of the task, with the Diverse Desire task as the easiest, and the Real-Apparent Emotion task as the most difficult. Participants will receive one point for each task passed successfully(range: 0-7). A higher score indicates a better ability of ToM.
Theory of mind (ToM) | 5 weeks, immediately after the intervention
  Children's ToM will be measured by the ToM scale developed by Wellman and Liu (2004). The seven-item scale was designed for the experimental to adminster in order according to the difficulty of the task, with the Diverse Desire task as the easiest, and the Real-Apparent Emotion task as the most difficult. Participants will receive one point for each task passed successfully (range: 0-7).A higher score indicates a better ability of ToM.
Working Memory Behavioural Manisfetation | 5 weeks, immediately after the intervention
  The Working Memory Subscale from the BRIEF-P is used to measure participants' daily behavioural manifestation of working memory reported by parents. The minimum raw score is 0 and maximum score is 17. A higher score indicates more severe deficits in working memory.
Working Memory Behavioural Manisfetation | before the intervention
  The Working Memory Subscale from the BRIEF-P is used to measure participants' daily behavioural manifestation of working memory reported by parents. The minimum raw score is 0 and maximum score is 17. A higher score indicates more severe deficits in working memory.

SECONDARY OUTCOMES:
ADHD symptoms(SNAP-IV) | before the intervention
  Swanson, Nolan and Pelham Parent Rating Scale (26 items, SNAP-IV; Chinese version; Gau et al., 2008) will be used to reflect the symptom severity of ADHD behaviors. The minimum raw score is 0 and maximum is 26. The higher score indicates a higher symptomatic presentation of ADHD behaviours.
ADHD symptoms(SNAP-IV) | 5 weeks, immediately after the intervention
  Swanson, Nolan and Pelham Parent Rating Scale (26 items, SNAP-IV; Chinese version; Gau et al., 2008) will be used to reflect the symptom severity of ADHD behaviors. The minimum raw score is 0 and maximum is 26. The higher score indicates a higher symptomatic presentation of ADHD behaviours.
Academic measures - Chinese word reading | before the intervention
  The Hong Kong Reading Ability Screening Test for Preschool Children (RAST-K) will be used to measure participants' Chinese word reading ability. The maximum score is 55 and the minimum is 0. The higher score indicates a better Chinese word reading ability.
Academic measures - Chinese word reading | 5 weeks, immediately after the intervention
  The Hong Kong Reading Ability Screening Test for Preschool Children (RAST-K) will be used to measure participants' Chinese word reading ability. The maximum score is 55 and the minimum is 0. The higher score indicates a better Chinese word reading ability.
Academic measures - English word reading | before the intervention
  An adapted English word reading assessment designed by the experimenters will be implemented to measure participants' English word reading ability. The maximum score is 55, and the minimum score is 0. A higher score indicates a higher ability of English word reading.
Academic measures - English word reading | 5 weeks, immediately after the intervention
  An adapted English word reading assessment designed by the experimenters will be implemented to measure participants' English word reading ability. The maximum score is 55, and the minimum score is 0. A higher score indicates a higher ability of English word reading.
Academic measures - Numeration | before the intervention
  The numeration subscale from Keymath-3 Diagnostic Assessment (Connolly, 2014) will be used to measure their number skills. The maximum score is 49 and the minimum score is 0. A higher score indicates a higher ability in numeration.
Academic measures - Numeration | 5 weeks, immediately after the intervention
  The numeration subscale from Keymath-3 Diagnostic Assessment (Connolly, 2014) will be used to measure their number skills. The maximum score is 49 and the minimum score is 0. A higher score indicates a higher ability in numeration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided